CLINICAL TRIAL: NCT00533689
Title: Study of the Long-Term Effect of Frequent Anti-VEGF Dosing on Retinal Function in Patients With Neovascular AMD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: TASMC-07-MG-209-CTIL
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Electrophysiology
MeSH Terms: interventions — Evoked Potentials, Visual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Electroretinography (ERG), Visual Evoked Potentials (VEP)

SUMMARY:
THis study aims to determine whether frequent dosing of intravitreal injections of Ranibizumab (Lucentis) or Bevacizumab (Avastin), which act as VEGF inhibitors, has a deleterious effect on the retina, studied by electrophysiologic testing.

This prospective, non-randomized clinical study will include patients assigned to intravitreal injection of Ranibizumab or Bevacizumab due to neovascular AMD. The patients will undergo repeat ophthalmic evaluation and intravitreal injections every 4-6 weeks, as long as will be deemed necessary. Periodic electrophysiologic evaluation including Electroretinogram (ERG), electro-oculogram (EOG) and Visual Evoked Potentials (VEP) tests will be performed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CNV secondary to AMD
* No other ocular disease
* No history of kerato-refractive surgery
* No epilepsy
* Ability to perform electrophysiologic study

Exclusion Criteria:

* Pregnancy
* Minority
* Epilepsy
* History of kerato-refractive surgery

Ages: 50 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 2008 (Estimated)
Dates: Start 2008-01; Study Completion 2010-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michaella Goldstein, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Anat Loewenstein, MD, Study Director — Tel-Aviv Sourasky Medical Center; Ido Perlman, PhD, Study Chair — Bruce Rappaport Faculty of Medicine, Technion, Haifa, Israel
Locations (1):
- Departent of Ophthalmlogy, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel